CLINICAL TRIAL: NCT05256186
Title: Effectiveness of Basketball Pre-injury Attack Program to Reduce the Susceptibility of Injury in Youth Basketball Players: a Randomized Controlled Trial
Brief Title: Effectiveness of Basketball Pre-injury Attack Program to Reduce the Susceptibility of Injury in Youth Basketball Players
Acronym: DPL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Associate Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123/2018 (phase 2)
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Injury;Sports; Biomechanical Lesions; Musculoskeletal Injury; Sports Physical Therapy
Keywords: Basketball; Prevention
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator
Masking Description: The study was blinded to the investigators who performed both recruitment and assessments. In this way, detection bias could be controlled. It was not possible to perform a double-blind study, since it was a physical intervention and the player knew that he/she was undergoing an intervention program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basketball pre-injury attack program (Experimental): The intervention group carried out a program for 24 weeks. The participant had to perform the program 3 days per week for 12-15' each day (training days with the team, prior to group activation).
  Interventions: Other: Basketball Pre-injury Attack program
- Control (No Intervention): The control group performed only the initial, follow-up (12 weeks) and final (24 weeks) evaluations.

INTERVENTIONS:
Other: Basketball Pre-injury Attack program — The intervention had a total duration of 24 weeks, with 3 sessions per week (before starting training) with a total duration of 12 to 15 minutes per session. Each session consisted of 8 exercises with a load of 2 to 3 series between 6 and 12 repetitions; and with a rest at the end of each series of <60 seconds.
  Arms: Basketball pre-injury attack program

SUMMARY:
Basketball is an impact, coordination-opposition sport with continuous contact among players and it is considered a sport of medium-high injury incidence. Players are force to have a physical condition appropriate to their practice and the demand to which they must respond due to the intensity of the efforts this sport requires. In order to achieve this, it is necessary to establish an evaluation protocol that allows the detection of functional deficiencies, to guide and conduct in a specific and early way every moment of players' health and growth.

The purpose of this study is to design, apply and analyze the effectiveness of a specific and individualized therapeutic exercise program (Basketball Pre-injury Attack) based on the approach of the functional deficiencies detected by the Basketball Injury Defense, to reduce the susceptibility to injury of youth basketball players (U14 - U17).

DETAILED DESCRIPTION:
The aim of this study is to design, apply and analyze the effectiveness of a specific and individualized therapeutic exercise program (Basketball Pre-injury Attack) based on the approach of functional deficiencies detected by the Basketball Injury Defense, to reduce the susceptibility to injury of training federated basketball players.

The specific objectives are:

To improve the deficiencies detected in mobility, stability, symmetry and jumping/landing technique of basketball players in training categories (U14, U16 and U17).

To structure and determine the contents of a specific and individualized therapeutic exercise program (Basketball Preinjury Attack) designed to improve the functional deficiencies of mobility, stability, symmetry and jumping/landing technique of training basketball players based on current scientific evidence.

To analyze whether adherence to the program is achieved by raising players' awareness of the importance and benefits of performing the exercises with correct technique.

To assess whether a decrease in the susceptibility to injury of training federated basketball players is achieved.

For this purpose, an experimental study was conducted as a single-blind, randomized, cluster-controlled clinical trial during the months of June 2019 to February 2020 (9 months). For the development of the methodology of this study, the guidelines of the CONSORT (Consolidated Standards of Reporting Trials) Statement were followed.

ELIGIBILITY:
Inclusion Criteria:

* Be between 10 and 17 years old
* Be an active player at the time of selection
* Sign the informed consent.

Exclusion Criteria:

* Being diagnosed with a psychological and/or psychiatric illness.
* Being diagnosed with an oncological disease.
* Be injured at the time of selection.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Ankle dorsiflexion under load | 1 year
  The Weight-bearing Lunge Test measured with the Leg Motion® system (Check Your Motion, Albacete) was used. Ankle dorsiflexion was recorded in centimeters.
Active hip, knee and ankle dorsiflexion | 1 year
  The Hurdle Step Test measured with the Leg Motion® system (Check Your Motion, Albacete) was used. A frontal and sagittal view was recorded with two filming devices so that the results could be analyzed later. Impairment was considered in those cases in which the subject was not able to step the foot over the rope during the hurdle step or if he/she performed adduction, internal or external rotation of the hip, and lost alignment between the hip, knee and ankle.
Ankle stability in monopodal loading | 1 year
  The Single Leg Squat Test was used and the criteria established by Perrot were used: it was considered stable if the foot remained in neutral position during the movement; and unstable if excessive pronation of the foot was evident during the movement or external rotation of the leg. To analyze the results, a frontal and sagittal view was recorded with two filming devices.
Monopodal dynamic knee valgus | 1 year
  The Single Leg Squat Test was used. The evaluator recorded a frontal and sagittal view with two filming devices. The knee was considered to be aligned if the patella was over the second toe.
Lumbo-pelvic stability | 1 year
  It was evaluated qualitatively with the Single Leg Squat Test and the Hurdle Step Test. To analyze the results, a frontal and sagittal view was recorded with two filming devices and the criteria established by Perrot were used. It was considered stable if there was minimal movement in all three planes, the pelvic girdle was aligned and there was no evidence of excessive anteroposterior tilt and/or trunk rotation. It was considered unstable if these criteria were not met.
Dynamic postural stability | 1 year
  It was analyzed qualitatively with the Single Leg Squat Test. The test was recorded with two filming devices (frontal and sagittal) and the criteria established by Perrot and Crossley were used. For this purpose, the deviation of the trunk with respect to the center of gravity was observed. It was considered stable if there was minimal translation of the center of mass, i.e., no lateral flexion/tilt, rotation or trunk flexion/extension.
Jumping/landing technique | 1 year
  It was analyzed with de Single Hop for distance Test. Ankle stability at landing, dynamic knee valgus, lumbopelvic stability and dynamic postural stability were analyzed.
Symmetry between the dominant and non-dominant limb | 1 year
  From the distance obtained in the Single Hop for distance Test, the Symmetry Index was calculated using the formula: (Distance dominant limb/Distance non-dominant limb)*100.

SECONDARY OUTCOMES:
Age | 1 year
  Recorded in years.
Category | 1 year
  According to the age of the participant could compete in 3 categories: U14, U16 or U17.
Gender | 1 year
  Female or male.
Weight | 1 year
  Weight was recorded in kg.
Height | 1 year
  Height was recorded in cm.
Body Mass Index (BMI) | 1 year
  It was calculated from the following formula [weight (kg) / height2 (m)].
Wingspan | 1 year
  The horizontal wingspan was recorded in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Adillón, MsC, Principal Investigator — University Rovira i Virgili
Locations (1):
- Federación Catalana de Baloncesto, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero Morales C, Calvo Lobo C, Rodriguez Sanz D, Sanz Corbalan I, Ruiz Ruiz B, Lopez Lopez D. The concurrent validity and reliability of the Leg Motion system for measuring ankle dorsiflexion range of motion in older adults. PeerJ. 2017 Jan 3;5:e2820. doi: 10.7717/peerj.2820. eCollection 2017. PMID 28070457
- [Background] Aerts I, Cumps E, Verhagen E, Wuyts B, Van De Gucht S, Meeusen R. The effect of a 3-month prevention program on the jump-landing technique in basketball: a randomized controlled trial. J Sport Rehabil. 2015 Feb;24(1):21-30. doi: 10.1123/jsr.2013-0099. Epub 2014 Jun 6. PMID 24911356
- [Background] Myer GD, Ford KR, McLean SG, Hewett TE. The effects of plyometric versus dynamic stabilization and balance training on lower extremity biomechanics. Am J Sports Med. 2006 Mar;34(3):445-55. doi: 10.1177/0363546505281241. Epub 2005 Nov 10. PMID 16282579
- [Background] Myklebust G, Engebretsen L, Braekken IH, Skjolberg A, Olsen OE, Bahr R. Prevention of anterior cruciate ligament injuries in female team handball players: a prospective intervention study over three seasons. Clin J Sport Med. 2003 Mar;13(2):71-8. doi: 10.1097/00042752-200303000-00002. PMID 12629423
- [Background] Moody JA, Naclerio F, Green P, Lloyd RS. Motor skill development in youths. En: Lloyd R, Oliver JL. Strength and Conditioning for Young Athletes: Science and Application. 1ª edición. New York:Routledge;2014
- [Background] Dill KE, Begalle RL, Frank BS, Zinder SM, Padua DA. Altered knee and ankle kinematics during squatting in those with limited weight-bearing-lunge ankle-dorsiflexion range of motion. J Athl Train. 2014 Nov-Dec;49(6):723-32. doi: 10.4085/1062-6050-49.3.29. PMID 25144599
- [Background] Baumbach SF, Braunstein M, Seeliger F, Borgmann L, Bocker W, Polzer H. Ankle dorsiflexion: what is normal? Development of a decision pathway for diagnosing impaired ankle dorsiflexion and M. gastrocnemius tightness. Arch Orthop Trauma Surg. 2016 Sep;136(9):1203-1211. doi: 10.1007/s00402-016-2513-x. Epub 2016 Jul 14. PMID 27418341
- [Background] Gonzalo-Skok O, Serna J, Rhea MR, Marin PJ. AGE DIFFERENCES IN MEASURES OF FUNCTIONAL MOVEMENT AND PERFORMANCE IN HIGHLY YOUTH BASKETBALL PLAYERS. Int J Sports Phys Ther. 2017 Oct;12(5):812-821. PMID 29181258
- [Background] Branta C, Haubenstricker J, Seefeldt V. Age changes in motor skills during childhood and adolescence. Exerc Sport Sci Rev. 1984;12:467-520. PMID 6734680
- [Background] Fort-Vanmeerhaeghe A, Gual G, Romero-Rodriguez D, Unnitha V. Lower Limb Neuromuscular Asymmetry in Volleyball and Basketball Players. J Hum Kinet. 2016 Apr 13;50:135-143. doi: 10.1515/hukin-2015-0150. eCollection 2016 Apr 1. PMID 28149351
- [Background] Doherty C, Delahunt E, Caulfield B, Hertel J, Ryan J, Bleakley C. The incidence and prevalence of ankle sprain injury: a systematic review and meta-analysis of prospective epidemiological studies. Sports Med. 2014 Jan;44(1):123-40. doi: 10.1007/s40279-013-0102-5. PMID 24105612
- [Background] McKeon PO, Hertel J. Systematic review of postural control and lateral ankle instability, part I: can deficits be detected with instrumented testing. J Athl Train. 2008 May-Jun;43(3):293-304. doi: 10.4085/1062-6050-43.3.293. PMID 18523566
- [Background] Perrott MA, Pizzari T, Opar M, Cook J. Development of clinical rating criteria for tests of lumbopelvic stability. Rehabil Res Pract. 2012;2012:803637. doi: 10.1155/2012/803637. Epub 2011 Dec 29. PMID 22263111
- [Background] Teyhen D, Bergeron MF, Deuster P, Baumgartner N, Beutler AI, de la Motte SJ, Jones BH, Lisman P, Padua DA, Pendergrass TL, Pyne SW, Schoomaker E, Sell TC, O'Connor F. Consortium for health and military performance and American College of Sports Medicine Summit: utility of functional movement assessment in identifying musculoskeletal injury risk. Curr Sports Med Rep. 2014 Jan-Feb;13(1):52-63. doi: 10.1249/JSR.0000000000000023. PMID 24412892
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287